CLINICAL TRIAL: NCT06269315
Title: Assessment of Skin Barrier Disruption Due to Daily Use of Cleaning Products and Hand Disinfectants
Acronym: SBDDCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Institute of Allergy and Asthma Research (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SBDDCP
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Control Condition (PBS); Household Detergent Exposure; Hand Disinfectant Exposure; Surfactant Exposure; Other Ingredients Exposure

STUDY DESIGN:
Intervention Model Description: 1. Skin Cleansing and Testing Patch Preparation:
     Prepare a test set of patch testing tapes, each containing a small amount of a different household cleaner, hand disinfectant, their ingredients, and control with proper dilution. The safety dose of the tested products and agents will be defined beforehand.
     Before exposure, selected areas of forearm skin will be cleaned and moistened. Electrical impedance will be measured by electrical impedance spectroscopy (EIS) to assess skin barrier integrity.
  2. Patch Application:
  Apply the prepared patches on the skin of the forearm. Patches will be removed after 5 minutes of exposure.
  During the exposure period, subjects will be instructed not to touch, wash, or wet the exposed area to avoid interfering with the action of the testing reagents. 3. Patch Removal and Post-Exposure Monitoring:
  The patch will be gently removed from the skin. Exposed areas of skin will be evaluated by EIS at specific times up to 24 hours after the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure arm (Experimental): Prepared test products, such as household cleaner, hand disinfectant, their ingredients, and control on patch testing tapes will be posted on the selected areas of forearm skin.
  Interventions: Other: Cleaning product exposure

INTERVENTIONS:
Other: Cleaning product exposure — Exposure of a small amount of a different household cleaner, hand disinfectant, their ingredients, and control with proper dilution on forearm of donors

SUMMARY:
The goal of this clinical trial is to assess the effects of household detergents and hand disinfectants on human skin barrier integrity among healthy adult volunteers.

The main questions it aims to answer are:

* How does exposure to household detergents and hand disinfectants impact skin barrier function?
* Are there differences in skin barrier disruption between various types of cleaning agents and disinfectants?

Participants will:

Undergo patch testing with controlled amounts of household detergents and hand disinfectants on a small area of their skin.

Be monitored for adverse reactions during and after exposure. Have their skin barrier integrity assessed using electrical impedance spectroscopy at multiple time points post-exposure.

If there is a comparison group:

Researchers will compare the effects of different types of cleaning agents, hand disinfectants, and their ingredients on skin barrier integrity to determine variations in their impact.

DETAILED DESCRIPTION:
1. Core Message:

   Understanding the effects of detergent and disinfectant exposure on skin barrier integrity is crucial for public health, particularly given their widespread use.
2. Supporting Information:

   Studies suggest an association between cleaning agents and skin barrier disruption. Skin barrier function can be assessed using various methods, including electrical impedance spectroscopy (EIS).
3. Key Points:

   Scientific Question: Investigate how household detergent, hand disinfectant, and their ingredients exposure affect skin barrier function.

   Proposed Intervention: Conduct controlled human skin exposure experiments with properly diluted household detergents, hand disinfectants, and their ingredients.

   Scientific Basis: Previous research indicates potential risks associated with cleaning agent exposure and validates EIS as a suitable assessment tool.
4. Objectives:

   Hypothesis: Household detergent and hand disinfectant exposure damage skin barrier integrity.

   Primary Objective: Demonstrate the effect of cleaning agent exposure on skin barrier function.
5. Study Population and Procedures:

   Inclusion criteria: Healthy adult volunteers aged 18-65. Exclusion criteria: Individuals with chronic skin conditions, allergies, or recent systemic therapy.

   Recruitment through ongoing processes and physician referrals. Informed consent emphasizing voluntary participation and the right to withdraw.
6. Statistics and Methodology:

   Sample size: 50 participants. Intervention: Participants will be exposed to controlled amounts of household detergents, hand disinfectants, and their ingredients.

   Assessment methods: EIS for skin barrier integrity evaluation. Statistical methods: Analysis using appropriate tests to detect significant differences.
7. Regulatory Aspects and Safety:

   Compliance with ethical guidelines and local regulations. Immediate reporting of adverse events and regular safety monitoring.
8. Quality Control and Data Protection:

   Measures include personnel training, SOPs, and data security protocols. Data is handled with discretion and stored securely.
9. Monitoring and Registration:

   Regular monitoring by research institutions (SIAF and UZH). This study will be registered with the Swiss National Clinical Trial Portal (SNCTP via BASEC) and ClinicalTrials.gov.
10. Funding / Publication / Declaration of Interest:

Funding from Swiss National Foundation (Prof. Cezmi Akdis) and SciBase. Commitment to transparency, open science, and conflict-free reporting. Multicentre collaboration between SIAF and Department of Dermatology, UZH.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of healthy adult volunteers; 1. age between18 and 65 years, 2. Generally healthy and able to provide written informed consent. The choice of healthy adult volunteers without pre-existing skin conditions on site or allergies against tested products is justified.

Exclusion Criteria:

1. Severe dermatitis, eczema, psoriasis, or other chronic skin conditions.
2. History of hypersensitivity or allergies to tested product ingredients.
3. Current or recent systemic therapy for a skin condition in the past six months.
4. Pregnant or breastfeeding individuals.
5. Use of investigational drugs or participation in another trial in the last 30 days.
6. History of skin cancer or malignancies in the study area.
7. Significant sunburn, open wounds, or active skin infections in the study area.
8. Any medical condition that, per the investigator, might compromise safety or confound results.
9. Inability to follow study instructions or attend required clinic visits.
10. Gender Balance: To ensure gender balance, efforts will be made to recruit an equal number of male and female participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Skin barrier evaluation | before the application (0), right after the removal (5 min), 1, 3, and 24 hours after the treatment
  We will measure skin barrier integrity by electrical impedance spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Institute of Allergy and Asthma Research, Davos, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No